CLINICAL TRIAL: NCT03712085
Title: Using fMRI and sEMG to Evaluate the Effects and Mechanism on Abdominal Acupuncture Combined With Upper Limb Rehabilitation Training on Brain Plasticity of Hemiplegic Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: YN2018HK03
Record Dates: First submitted 2018-07-07; First posted 2018-10-19 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Brain Ischemia; Hemiplegic Patients With Stroke; Image Science; Electrophysiology of Neuromuscular; Abdominal Acupuncture
Keywords: Functional magnetic resonance imaging（fMRI）; Surface electromyography （sEMG）; Abdominal acupuncture; Brain Plasticity; Effects and mechanism
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group A (Active Comparator): Abdominal acupuncture and upper limb rehabilitation training
  Interventions: Other: Abdominal acupuncture
- Treatment Group B (Sham Comparator): Sham abdominal acupuncture and upper limb rehabilitation training
  Interventions: Other: Sham abdominal acupuncture
- Control Group (No Intervention): Upper limb rehabilitation only

INTERVENTIONS:
Other: Abdominal acupuncture — Abdominal acupuncture treatment method: 1.Acupoints selection :Zhongwan,Xiawan,Shangqu,Qihai,Guanyuan,Huaroumen,Upper rheumatic and Upper rheumatic external points etc.(Acupoints selection referred to Abdominal Acupuncture Therapy written by Bo Zhiyun ,the founder of Abdominal Acupuncture. 2.Treatment Duration: 30 minutes a session, once a day, 5 times a week for 3 weeks.
  Arms: Treatment Group A
Other: Sham abdominal acupuncture — Sham abdominal acupuncture Abdominal acupuncture treatment method: 1.Acupoints selection and treatment duration are the same as abdominal acupuncture. 3.Method：Using the sham abdominal acupuncture needles were produced by DONGBANG AcuPrime Acupuncture Instrument Co., Ltd. ( U.K.)The tip of the needle was exposed to 1mm of the cannula. The acupoint skin of patients was touched gently by the tip, and the tip of needle was lifted and removed from acupoint skin after 30s. Rest for 30 seconds ,then repeated 6 times, a total time of stimulation is 6min.
  Other Names: Upper limb rehabilitation training
  Arms: Treatment Group B

SUMMARY:
Using random number method to categorize the selected first onset patients with stroke who meet the inclusion criteria into 3 groups.The patients were randomly divided into treatment group A(abdominal acupuncture+upper limb rehabilitation training, 22 cases), treatment group B(Sham abdominal acupuncture+upper limb rehabilitation training, 22 cases),and control group(upper limb rehabilitation training, 22 cases). SEMG and fMRI examination and related stroke rehabilitation assessment scales were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. First onset stroke, Left hemiplegia, Right-handed，and diagnosed by brain CT or MRI;
2. Age 35 to 75 years old;
3. Course of disease 0.5 to 3 months with stable vital signs;
4. No cognitive impairment. Can understand and execute commands. MMSE score more than 7 points. ;
5. Can control the sitting balance. Brunnstrom stage of hemiplegic upper limb and hand is Ⅳ or V ，Fugl-Meyer Motor Assessment score of upper limb 20-50 point;
6. Agree to sign the informed consent;
7. Unilateral neglect.

Exclusion Criteria:

1. Recurrent stroke，subarachnoid hemorrhage, brain tumors patients;
2. Contraindication to undergo a 3T MR imaging;
3. Claustrophobia;
4. Have severe heart, hepatic or renal failure;
5. Don' t cooperate with the treatment;
6. Have participated in other clinical trails recently.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The integrity of the corticospinal tract | Diffusion tensor imaging(DTI) will be tested before treatment and 4 weeks after treatment,twice totally.
  The integrity of the corticospinal tract will be tested by diffusion trnsor imaging(DTI) of craniocerebral functional magnetic resonance imaging examination using magetic angiography to measure the changes caused by neuronal activity.We will observe the shape and integrity of the corticospinal tract.
Motor function of muscles | SEMG will be tested before and after 4 weeks treatment,twice totally.
  Common measures of sEMG will be tested. See the study protocol for details.

SECONDARY OUTCOMES:
Wolf Motor Function Test | Before treatment, 2 weeks and 4 weeks after treatment， 3 times totally.
  See the study protocol for details
Brunnstrom staging of upper limb movement | Before treatment, 2 weeks and 4 weeks after treatment， 3 times totally.
  See the study protocol for details
Fugl-Meyer Motor Assessment of upper limb | Before treatment, 2 weeks and 4 weeks after treatment， 3 times totally.
  See the study protocol for details
Modified Barthel Index，MBI | Before treatment, 2 weeks and 4 weeks after treatment， 3 times totally.
  See the study protocol for details

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Chen, Master, Principal Investigator — Director of the rehabilitation department; Vincet Chi-kwan Cheung, Doctor, Principal Investigator — Assistant professor
Locations (2):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Informed Consent Form (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03712085/ICF_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03712085/SAP_001.pdf
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03712085/Prot_002.pdf